CLINICAL TRIAL: NCT03033368
Title: Treatment Switch From Efavirenz to Rilpivirine in Virologically-suppressed HIV-infected Thai Adolescents
Brief Title: Rilpivirine in Virologically Suppressed Adolescents
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPV
Record Dates: First submitted 2016-10-22; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: immunological outcome; virologic outcomes; HIV-1 infected adolescents; EFV switch to RPV; Rilpivirine pharmacokinetic; neuropsychiatric adverse events
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- opened label (Experimental): Open-label, single-arm study, rilpivirine is the study drug
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Rilpivirine — Rilpivirine 25 mg tablet
  Other Names: Edurant

SUMMARY:
To describe the immunologic and virologic outcomes (HIV RNA, CD4) following switching from EFV to RPV in virologically suppressed adolescents

DETAILED DESCRIPTION:
Study Procedures:

At screening, the informed consent process will be provided to participant, or participant legally acceptable representatives before any study procedure. Only adolescents who know their HIV status will be asked to give assent.

Twenty adolescents followed at HIV-NAT and the Department of Pediatrics, Faculty of Medicine, Chulalongkorn University will be asked to participate in the PK sub study. Participant who are enrolled in the PK substudy will be asked to take RPV in the morning after breakfast and then commence the PK evaluations after this witnessed dose. After the PK study at week 4, Participant will be followed with the other 80 adolescents until the end of the study. Participant will be asked to provide a small hair sample for RPV concentrations at weeks 4, 12, 24, and 48 after switching. This is an option therefore participant can refuse to provide their hair samples at any visits. HIV RNA levels will be performed at baseline, week 12, 24 and 48 visits. If the HIV-RNA at any visits is between >50 copies/ml, the HIV-RNA test will be repeated within 4-8 weeks with adherence improvement counseling. At any visit, if HIV-RNA is ≥1000 copies/ml, genotypic resistance testing will be performed. Modification of treatment both for resistance and safety consideration will be subject to the site principal investigator's decision.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adolescents aged 12-18 years;
* Body weight >25 kilograms;
* Currently treated with stable EFV-based HAART (EFV plus two nucleoside or nucleotide reverse transcriptase inhibitors [N(t)RTI]) for >3 months prior to enrollment;
* Plasma HIV RNA <50 copies/ml within the last 12 months;
* ALT <200 IU/L within the last 12 months;
* Caregivers give written informed consent and adolescents who know their HIV status (i.e., have been fully disclosed to) give assent

Exclusion Criteria:

* Has evidence of NNRTI-associated resistance mutation(s) from previous genotypic resistance testing;
* Currently has PI(s) in the HAART regimen;
* Has currently active HIV-related infection(s), (The subject can be enrolled after the infection is under controlled);
* Has significant medical problem(s) that would compromise study results (in the site principal investigator's opinion);
* Pregnancy (postpartum women are allowed);
* Concomitant treatment with drugs known to effect the PK of RPV (carbamazepine, phenobarbital, phenytoin, rifampicin, rifabutin, omeprazole, esomeprazole, lansoprazole, erythromycin, clarithromycin, azithromycin, roxithromycin)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of adolescents with HIV-RNA <50 copies/ml at 48 weeks after switching. | 48 weeks

SECONDARY OUTCOMES:
Change in neuropsychiatric test scores | Baseline and week 24
  Using Trail Making Test and Coding subtest of WISC-III Wisconsin Card Sorting Test (WCST) Non-verbal part of Standard Progressive Matrices
Change in quality of life (QOL) score | Baseline, week 4 and week 24
  Using PedsQLTM 4.0
Change in lipid profiles after switching to RPV-containing regimens | Baseline, week 24, and week 48
  Measure cholesterol (mg/dl), LDL (mg/dl), HDL (mg/dl), triglyceride (mg/dl)
Change in fasting blood sugar after switching to RPV-containing regime | Baseline, week 24, and week 48
  Measue fasting blood sugar (mg/dl)
Intensive PK parameter (Area under the plasma concentration-time curve; AUC0-24) of RPV in 20 subjects at 4 weeks after switching to RPV-containing regimens. | week 4
  Measure area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24): unit; ng.h/ml
Intensive PK parameter (maximum observed concentration of drug in plasma ;(Cmax) ) of RPV in 20 subjects at 4 weeks after switching to RPV-containing regimens. | week 4
  Measue maximum observed concentration of drug in plasma (Cmax) : unit; ng/ml
Intensive PK parameter (Minimum concentration of drug in plasma; (Ctrough)) of RPV in 20 subjects at 4 weeks after switching to RPV-containing regimens. | week 4
  Measure minimum concentration of drug in plasma (Ctrough) : unit; ng/ml
Description of resistance mutations in the adolescents with RPV treatment failure | baseline, week 12, week 24 and week 48
  At any visit, if HIV-RNA is ≥1000 copies/ml, genotypic resistance testing will be performed. Using HIV-1 Antiretroviral drug resistance ViriSeq HIV-1 genotyping

IPD SHARING:
Plan to Share IPD: Yes
Investigator plan to the clinical data

REFERENCES:
- [Derived] Jantarabenjakul W, Anugulruengkitt S, Kasipong N, Thammajaruk N, Sophonphan J, Bunupuradah T, Cressey TR, Colbers A, Burger DM, Phongsamart W, Puthanakit T, Pancharoen C; HIVNAT 220 study. Pharmacokinetics of rilpivirine and 24-week outcomes after switching from efavirenz in virologically suppressed HIV-1-infected adolescents. Antivir Ther. 2018;23(3):259-265. doi: 10.3851/IMP3198. PMID 28994660